CLINICAL TRIAL: NCT06130735
Title: Computerized Cognitive Training: Characterization of Factors That Predict Cognitive Enhancement in Acquired Brain Injury
Brief Title: Impact of Intensive Computerized Cognitive Training
Acronym: CCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Fujifilm (Industry)
Responsible Party: Principal Investigator, Kirk Daffner, MD, Chief, Division of Cognitive and Behavioral Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P003401
Record Dates: First submitted 2023-10-30; First posted 2023-11-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Acquired Brain Injury; Mild Cognitive Impairment; Mild Neurocognitive Disorder
Keywords: computerized cognitive training; working memory; acquired brain injury; mild neurocognitive impairment; neuropsychological testing; BDNF; event-related potentials
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Cognitive Training (Experimental): See section of intervention/treatment for additional information.
  Interventions: Behavioral: Cognitive Computerized Training

INTERVENTIONS:
Behavioral: Cognitive Computerized Training — Participants will log into ABI Wellness Platform five days per week (M-T-W-Th-F) and train using the Symbol Relations module for 45 to 60 minutes. Every other week, participants will meet with their training facilitator via zoom to review training progress and troubleshoot any training-related questions.

SUMMARY:
To investigate factors that predict cognitive enhancement following engagement in an intensive Computerized Cognitive Training Protocol.

DETAILED DESCRIPTION:
To investigate factors that predict cognitive enhancement following engagement in an intensive 6-month, 5 days per week training use the ABI Wellness BEARS platform and Brainex Software Symbol Relations Module.

The study will examine the impact of intensive working memory training on neurocognitive markers of brain plasticity (intervention-related changes) in 1) performance on neuropsychological tests, 2) BDNF levels in blood and salivary, 3) ERP measures of working memory, and 4) resting state fMRI and structural MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Mass General Brigham Health System with primary attention and executive functioning difficulties and/or a diagnosis of mild cognitive disorder or mild neurocognitive disorder (non-amnestic profile), due to an acquired brain injury (ABI) sustained at least 12 months prior to study contact.
* Ages 25-65 years old
* Proficiency in English
* Willing and able to complete all study-related activities for 12 months, including travel to Brigham and Women's Hospital (Boston) for four in-person assessment visits and two serum and saliva sample collections.
* Access to a computer with webcam and stable internet.
* A reliable study informant who can complete one questionnaire about participant's cognition/daily functioning, at four time points.

Exclusion Criteria:

* History of alcohol or substance abuse, or dependence, within the past 2 years, as per DSM-5 criteria.
* High likelihood of an underlying progressive neurodegenerative disorder.
* Evidence of moderate to severe cognitive disorder, based on a score of 21 or less on the Mini-Mental Status Examination (MMSE) (Tombaugh & McIntyre, 1992).
* Patient Health Questionnaire (PHQ)-9 (Kroenke et al., 2010) Score ≥ 19, unless deemed by treating provider not to have active depression (e.g., adjustment disorder, grief reaction).
* Active psychotic symptoms.
* Severe sensory losses such that participants would unlikely be able to participate in the study training, even with substantial accommodations (self-report of extreme difficulty reading ordinary newspaper print or a performance-tested corrected vision test score of worse than 20/30).
* Communication difficulties that prevent the participant from effectively participating in this highly interactive study protocol (based on interviewer's rating of a person's ability to be understood and to understand others).
* Current participation in a pharmacological, or other interventional research trial.
* Life expectancy of < 2 years.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive outcome measures | 6 months
  We will use age-corrected standard scores of the NIH toolbox Total Cognitive Composite, Fluid Intelligence Composite, and individual scores on RAVLT, Verbal Fluency, and Trailmaking Task as cognitive outcome measures.
Changes in BDNF Levels in blood and saliva | 6 months
  Using FUJIFILM high sensitivity ELISA kits and commercially available ELISA kits.

SECONDARY OUTCOMES:
Self-report exercise and physical activity | 6 months
  Physical Activity Scale for the Elderly (questionnaire).
  Measures walking, moderate, and vigorous activity. Zero lower limit, no upper limit. Higher values indicate more physical activity.
Intervention-related changes in ERP measures, such as the P3 component (P3a and P3b) | 6 months
  1) Measured in response to verbal and visual working memory tasks
Intervention-related changes in resting state fMRI | 6 months
  A group ICA analysis procedure will be applied to pre- and post-intervention rs-fMRI BOLD signal activity. Correlations will be explored between fMRI parameters, cognitive, and training data (e.g NIH toolbox Total Cognitive Composite, Fluid Intelligence Composite, Crystallized Composite, CCT engagement and progress).
Quality of life self-report | 6 months
  Flanagan Quality of Life Scale (questionnaire).
  Measures quality of life. Likert scale 0-112, higher values indicate higher quality of life.
Sleep | 6 months
  Medical Outcomes Study Sleep Scale (questionnaire)
  Likert scale measuring sleep quality and sleep problems index. 0-60 with greater values representing higher sleep quality and lower sleep problems.
Anxiety | 6 months
  Generalized Anxiety Disorder 7 Item Scale (questionnaire)
  Likert scale measuring severity of anxiety. 0-21 with greater values representing more severe anxiety.
Depression | 6 months
  Patient Health Questionnaire Depression Scale (questionnaire)
  Likert scale measuring the severity of depression. 0-24 with higher scores representing more severe depression.
Self-report on impact of fatigue | 6 months
  Modified Fatigue Impact Scale
  Likert scale on the impact of fatigue on one's physical, cognitive, and psychosocial activity. 0-84 with higher scores indicating a greater impact of fatigue on a person's activities.
Feelings about cognitive/thinking skills | 6 months
  Cognitive Self- Efficacy Questionnaire
  Likert scale on feelings people have about their cognition/thinking skills. 0-72 with a higher score indicating more positive feelings regarding the efficacy of ones cognitive/thinking abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Kim C Willment, PhD, Principal Investigator — Brigham and Women's Hospital; Kirk R Daffner, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norman A, Curro V, Holloway M, Percuklievska N, Ferrario H. Experiences of individuals with acquired brain injury and their families interacting with community services: a systematic scoping review. Disabil Rehabil. 2023 Feb;45(4):739-751. doi: 10.1080/09638288.2022.2043465. Epub 2022 Mar 4. PMID 35244507
- [Background] Amariglio RE, Donohue MC, Marshall GA, Rentz DM, Salmon DP, Ferris SH, Karantzoulis S, Aisen PS, Sperling RA; Alzheimer's Disease Cooperative Study. Tracking early decline in cognitive function in older individuals at risk for Alzheimer disease dementia: the Alzheimer's Disease Cooperative Study Cognitive Function Instrument. JAMA Neurol. 2015 Apr;72(4):446-54. doi: 10.1001/jamaneurol.2014.3375. PMID 25706191
- [Background] Billig AR, Feng NC, Behforuzi H, McFeeley BM, Nicastri CM, Daffner KR. Capacity-limited resources are used for managing sensory degradation and cognitive demands: Implications for age-related cognitive decline and dementia. Cortex. 2020 Dec;133:277-294. doi: 10.1016/j.cortex.2020.09.005. Epub 2020 Sep 24. PMID 33157347
- [Background] Biswal BB. Resting state fMRI: a personal history. Neuroimage. 2012 Aug 15;62(2):938-44. doi: 10.1016/j.neuroimage.2012.01.090. Epub 2012 Jan 24. PMID 22326802
- [Background] Buckner RL, Krienen FM, Yeo BT. Opportunities and limitations of intrinsic functional connectivity MRI. Nat Neurosci. 2013 Jul;16(7):832-7. doi: 10.1038/nn.3423. Epub 2013 Jun 25. PMID 23799476
- [Background] Burckhardt CS, Anderson KL, Archenholtz B, Hagg O. The Flanagan Quality Of Life Scale: evidence of construct validity. Health Qual Life Outcomes. 2003 Oct 23;1:59. doi: 10.1186/1477-7525-1-59. PMID 14613563
- [Background] Chen K, Azeez A, Chen DY, Biswal BB. Resting-State Functional Connectivity: Signal Origins and Analytic Methods. Neuroimaging Clin N Am. 2020 Feb;30(1):15-23. doi: 10.1016/j.nic.2019.09.012. PMID 31759568
- [Background] Coulter CL, Weber JM, Scarvell JM. Group physiotherapy provides similar outcomes for participants after joint replacement surgery as 1-to-1 physiotherapy: a sequential cohort study. Arch Phys Med Rehabil. 2009 Oct;90(10):1727-33. doi: 10.1016/j.apmr.2009.04.019. PMID 19801063
- [Background] Daffner KR, Chong H, Sun X, Tarbi EC, Riis JL, McGinnis SM, Holcomb PJ. Mechanisms underlying age- and performance-related differences in working memory. J Cogn Neurosci. 2011 Jun;23(6):1298-314. doi: 10.1162/jocn.2010.21540. Epub 2010 Jul 9. PMID 20617886
- [Background] Kersel DA, Marsh NV, Havill JH, Sleigh JW. Neuropsychological functioning during the year following severe traumatic brain injury. Brain Inj. 2001 Apr;15(4):283-96. doi: 10.1080/02699050010005887. PMID 11299130
- [Background] Denboer JW, Nicholls C, Corte C, Chestnut K. National Institutes of Health Toolbox Cognition Battery. Archives of Clinical Neuropsychology. 2014; 29(7): 692-694
- [Background] Hays RD, Stewart AL. Measuring functioning and well-being: The Medical Outcomes Study Approach. Duke University Press. 1992.
- [Background] Holloway M, Tasker R. The Experiences of Relatives of People with Acquired Brain Injury (ABI) of the Condition and Associated Social and Health Care Services. Journal of Long-term Care. 2019, p.99-110
- [Background] Ivnik RJ, Malec JF, Smith GE, Tangalos EG, Petersen, RC. Neuropsychological tests' norms above age 55: COWAT, BNT, MAE Token, WRAT-R Reading, AMNART, STROOP, TMT, and JLO. The Clinical Neuropsychologist. 1996; 10(3): 262-278.
- [Background] Jones JM, Haslam SA, Jetten J, Williams WH, Morris R, Saroyan S. That which doesn't kill us can make us stronger (and more satisfied with life): the contribution of personal and social changes to well-being after acquired brain injury. Psychol Health. 2011 Mar;26(3):353-69. doi: 10.1080/08870440903440699. PMID 20419563
- [Background] Kersel DA, Marsh NV, Havill JH, Sleigh JW. Psychosocial functioning during the year following severe traumatic brain injury. Brain Inj. 2001 Aug;15(8):683-96. doi: 10.1080/02699050010013662. PMID 11485609
- [Background] Kurasik S. Group dynamics in the rehabilitation of hemiplegic patients. J Am Geriatr Soc. 1967 Sep;15(9):852-5. doi: 10.1111/j.1532-5415.1967.tb02443.x. No abstract available. PMID 5341016
- [Background] Ledreux A, Hakansson K, Carlsson R, Kidane M, Columbo L, Terjestam Y, Ryan E, Tusch E, Winblad B, Daffner K, Granholm AC, Mohammed AKH. Differential Effects of Physical Exercise, Cognitive Training, and Mindfulness Practice on Serum BDNF Levels in Healthy Older Adults: A Randomized Controlled Intervention Study. J Alzheimers Dis. 2019;71(4):1245-1261. doi: 10.3233/JAD-190756. PMID 31498125
- [Background] Levin C, Chisholm D.
- [Background] Lezak MD, Howieson DB, Bigler ED, & Tranel D. Neuropsychological assessment, 5th ed. APA PsychNet. 2012.
- [Background] Nicastri CM, McFeeley BM, Simon SS, Ledreux A, Hakansson K, Granholm AC, Mohammed AH, Daffner KR. BDNF mediates improvement in cognitive performance after computerized cognitive training in healthy older adults. Alzheimers Dement (N Y). 2022 Aug 30;8(1):e12337. doi: 10.1002/trc2.12337. eCollection 2022. PMID 36089933
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Porter S, Torres IJ, Panenka W, Rajwani Z, Fawcett D, Hyder A, Virji-Babul N. Changes in brain-behavior relationships following a 3-month pilot cognitive intervention program for adults with traumatic brain injury. Heliyon. 2017 Aug 4;3(8):e00373. doi: 10.1016/j.heliyon.2017.e00373. eCollection 2017 Aug. PMID 28795168
- [Background] Retan R, Wolfson D. The Halstead-Reitan neuropsychological test battery: Theory and clinical interpretation. Neuropsychology Press. 1985.
- [Background] Rosazza C, Minati L. Resting-state brain networks: literature review and clinical applications. Neurol Sci. 2011 Oct;32(5):773-85. doi: 10.1007/s10072-011-0636-y. Epub 2011 Jun 11. PMID 21667095
- [Background] Schulenberg SE, Yutrzenka BA, Gohm CL. The Computer Aversion, Attitudes, and Familiarity Index (CAAFI): A Measure for the Study of Computer-Related Constructs. Journal of Educational Computing Research. 2006; 34(2): 129-146.
- [Background] Sevick et al. Alterations in Resting State Functional Connectivity in Patients with Traumatic Brain Injury Following a 3-month Pilot Cognitive Intervention Program. Poster Presented at: UBC Department of Psychiatry 2020 Virtual Research Day. 2020.
- [Background] Simon SS, Tusch ES, Feng NC, Hakansson K, Mohammed AH, Daffner KR. Is Computerized Working Memory Training Effective in Healthy Older Adults? Evidence from a Multi-Site, Randomized Controlled Trial. J Alzheimers Dis. 2018;65(3):931-949. doi: 10.3233/JAD-180455. PMID 30103334
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Tennstedt SL, Unverzagt FW. The ACTIVE study: study overview and major findings. J Aging Health. 2013 Dec;25(8 Suppl):3S-20S. doi: 10.1177/0898264313518133. No abstract available. PMID 24385638
- [Background] Tombaugh TN, McIntyre NJ. The mini-mental state examination: a comprehensive review. J Am Geriatr Soc. 1992 Sep;40(9):922-35. doi: 10.1111/j.1532-5415.1992.tb01992.x. PMID 1512391
- [Background] Trahey PJ. A comparison of the cost-effectiveness of two types of occupational therapy services. Am J Occup Ther. 1991 May;45(5):397-400. doi: 10.5014/ajot.45.5.397. PMID 1904685
- [Background] Troyer AK, Leach L, Vandermorris S, Rich JB. The measurement of participant-reported memory across diverse populations and settings: a systematic review and meta-analysis of the Multifactorial Memory Questionnaire. Memory. 2019 Aug;27(7):931-942. doi: 10.1080/09658211.2019.1608255. Epub 2019 Apr 25. PMID 31020904
- [Background] Tulsky DS, Kisala PA. Overview of the Spinal Cord Injury-Functional Index (SCI-FI): Structure and Recent Advances. Arch Phys Med Rehabil. 2022 Feb;103(2):185-190. doi: 10.1016/j.apmr.2021.10.006. Epub 2021 Oct 28. PMID 34756875
- [Background] Tusch ES, Alperin BR, Ryan E, Holcomb PJ, Mohammed AH, Daffner KR. Changes in Neural Activity Underlying Working Memory after Computerized Cognitive Training in Older Adults. Front Aging Neurosci. 2016 Nov 8;8:255. doi: 10.3389/fnagi.2016.00255. eCollection 2016. PMID 27877122
- [Background] Vakil E, Blachstein H. Rey Auditory-Verbal Learning Test: structure analysis. J Clin Psychol. 1993 Nov;49(6):883-90. doi: 10.1002/1097-4679(199311)49:63.0.co;2-6. PMID 8300877
- [Background] Vos T, Corry J, Haby MM, Carter R, Andrews G. Cost-effectiveness of cognitive-behavioural therapy and drug interventions for major depression. Aust N Z J Psychiatry. 2005 Aug;39(8):683-92. doi: 10.1080/j.1440-1614.2005.01652.x. PMID 16050922
- [Background] Walsh RS, Fortune DG, Gallagher S, Muldoon OT. Acquired brain injury: combining social psychological and neuropsychological perspectives. Health Psychol Rev. 2014;8(4):458-72. doi: 10.1080/17437199.2012.733914. Epub 2012 Oct 22. PMID 25211210
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Wechsler D. Manual for the Wechsler Adult Intelligence Scale. Psychological Corporation. 1955.
- [Background] Zanca JM, Dijkers MP, Hsieh CH, Heinemann AW, Horn SD, Smout RJ, Backus D. Group therapy utilization in inpatient spinal cord injury rehabilitation. Arch Phys Med Rehabil. 2013 Apr;94(4 Suppl):S145-53. doi: 10.1016/j.apmr.2012.11.049. PMID 23527770
- See also: Experiences of individuals with acquired brain injury and their families interacting with community services: a systematic scoping review — https://pubmed.ncbi.nlm.nih.gov/35244507/
- See also: Tracking early decline in cognitive function in older individuals at risk for Alzheimer's disease dementia: the Alzheimer's Disease Cooperative Study Cognitive Function Instrument — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4397164/
- See also: Capacity-limited resources are used for managing sensory degradation and cognitive demands: Implications for age-related cognitive decline and dementia — https://pubmed.ncbi.nlm.nih.gov/33157347/
- See also: Resting state fMRI: a personal history — https://pubmed.ncbi.nlm.nih.gov/22326802/
- See also: Opportunities and limitations of intrinsic functional connectivity MRI — https://pubmed.ncbi.nlm.nih.gov/23799476/
- See also: The Flanagan Quality Of Life Scale: evidence of construct validity — https://pubmed.ncbi.nlm.nih.gov/14613563/
- See also: Resting-State Functional Connectivity: Signal Origins and Analytic Methods — https://pubmed.ncbi.nlm.nih.gov/31759568/
- See also: Group physiotherapy provides similar outcomes for participants after joint replacement surgery as 1-to-1 physiotherapy: a sequential cohort study — https://pubmed.ncbi.nlm.nih.gov/19801063/
- See also: Mechanisms Underlying Age- and Performance-related Differences in Working Memory — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3076134/
- See also: National Institutes of Health Toolbox Cognition Battery — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4263919/
- See also: Neuropsychological functioning during the year following severe traumatic brain injury — https://pubmed.ncbi.nlm.nih.gov/11299130/
- See also: The Experiences of Relatives of People with Acquired Brain Injury (ABI) of the Condition and Associated Social and Health Care Services — https://journal.ilpnetwork.org/articles/10.31389/jltc.20
- See also: That which doesn't kill us can make us stronger (and more satisfied with life): the contribution of personal and social changes to well-being after acquired brain injury — https://pubmed.ncbi.nlm.nih.gov/20419563/
- See also: Psychosocial functioning during the year following severe traumatic brain injury — https://pubmed.ncbi.nlm.nih.gov/11485609/
- See also: Group dynamics in the rehabilitation of hemiplegic patients — https://pubmed.ncbi.nlm.nih.gov/5341016/
- See also: Differential Effects of Physical Exercise, Cognitive Training, and Mindfulness Practice on Serum BDNF Levels in Healthy Older Adults: A Randomized Controlled Intervention Study — https://pubmed.ncbi.nlm.nih.gov/31498125/
- See also: BDNF mediates improvement in cognitive performance after computerized cognitive training in healthy older adults — https://pubmed.ncbi.nlm.nih.gov/36089933/
- See also: The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review — https://pubmed.ncbi.nlm.nih.gov/20633738/
- See also: Modified Fatigue Impact Scale — https://www.sralab.org/rehabilitation-measures/modified-fatigue-impact-scale
- See also: Changes in brain-behavior relationships following a 3-month pilot cognitive intervention program for adults with traumatic brain injury — https://pubmed.ncbi.nlm.nih.gov/28795168/
- See also: Resting-state brain networks: literature review and clinical applications — https://pubmed.ncbi.nlm.nih.gov/21667095/
- See also: Is Computerized Working Memory Training Effective in Healthy Older Adults? Evidence from a Multi-Site, Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/30103334/
- See also: The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue — https://pubmed.ncbi.nlm.nih.gov/7636775/
- See also: The ACTIVE study: study overview and major findings — https://pubmed.ncbi.nlm.nih.gov/24385638/
- See also: The mini-mental state examination: a comprehensive review — https://pubmed.ncbi.nlm.nih.gov/1512391/
- See also: A comparison of the cost-effectiveness of two types of occupational therapy services — https://pubmed.ncbi.nlm.nih.gov/1904685/
- See also: The measurement of participant-reported memory across diverse populations and settings: a systematic review and meta-analysis of the Multifactorial Memory Questionnaire — https://pubmed.ncbi.nlm.nih.gov/31020904/
- See also: Overview of the Spinal Cord Injury-Functional Index (SCI-FI): Structure and Recent Advances — https://pubmed.ncbi.nlm.nih.gov/34756875/
- See also: Changes in Neural Activity Underlying Working Memory after Computerized Cognitive Training in Older Adults — https://pubmed.ncbi.nlm.nih.gov/27877122/
- See also: Rey Auditory-Verbal Learning Test: structure analysis — https://pubmed.ncbi.nlm.nih.gov/8300877/
- See also: Cost-effectiveness of cognitive-behavioural therapy and drug interventions for major depression — https://pubmed.ncbi.nlm.nih.gov/16050922/
- See also: Acquired brain injury: combining social psychological and neuropsychological perspectives — https://pubmed.ncbi.nlm.nih.gov/25211210/
- See also: The Physical Activity Scale for the Elderly (PASE): development and evaluation — https://pubmed.ncbi.nlm.nih.gov/8437031/
- See also: Group therapy utilization in inpatient spinal cord injury rehabilitation — https://pubmed.ncbi.nlm.nih.gov/23527770/